CLINICAL TRIAL: NCT06953154
Title: Monocyte Distribution Width (MDW): An Early Marker of Sepsis in Patients With Comorbidities
Acronym: MDW
Status: Completed | Type: Observational
Sponsor: Hôpital Universitaire Sahloul (Other)
Responsible Party: Principal Investigator, Riadh Boukef, service chief, Hôpital Universitaire Sahloul
Other Study IDs: Emergency Department
Record Dates: First submitted 2025-03-07; First posted 2025-05-01 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: monocyte distribution width — We compare the measured value with the MDW threshold value already established in the literature and its correlation with the SOFA score, qSOFA, lactate, and PVI in terms of sensitivity, specificity, negative predictive value (NPV), and positive predictive value (PPV).

SUMMARY:
In patients with the aforementioned comorbidities, septic conditions are common and associated with high mortality rates. Early diagnosis, along with prompt and appropriate management, has become a major challenge for emergency departments. However, it is often difficult to determine whether sepsis is the primary factor behind clinical decompensation, especially in patients with complex comorbidities where symptoms may be nonspecific and overlap with other causes of deterioration. This diagnostic uncertainty complicates the timely initiation of targeted treatment, making the role of biomarkers even more crucial.

The measurement of sepsis biomarkers is widely used in clinical practice to enhance diagnostic accuracy, but there remains a need for a more reliable biomarker. A biomarker with higher sensitivity and negative predictive value (NPV) is essential for the early initiation of treatment. Several European and American studies have demonstrated the added value of MDW as an early predictor of sepsis in patients admitted to intensive care units, as well as its diagnostic performance when combined with the qSOFA score.

In the literature, the MDW threshold is established at 21.5, offering optimal diagnostic power with good sensitivity and specificity, supporting its clinical application and its approval by the United States Food and Drug Administration (FDA) and the European Conformity (CE).

In Tunisia, few studies have focused on the effectiveness of this non-invasive tool in septic patients in emergency settings and its reliability in this context, highlighting the relevance of our research.

DETAILED DESCRIPTION:
We will test the effectiveness of MDW in the early diagnosis of sepsis as a factor of decompensation in patients with comorbidities: renal failure, heart failure, and COPD.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years admitted to the emergency department for decompensation of congestive heart failure or renal failure, or exacerbation of COPD.

Exclusion Criteria:

* Patients who received antibiotic treatment in the past 7 days, pregnant women, children, non-consenting patients, patients with a history of malignant hematologic disease, polytransfused patients or those who recently received a transfusion, and patients whose MDW was not reported due to ineffective monocyte counting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with comorbidities (heart failure , renal failure and COPD)
Sampling Method: Probability Sample
Enrollment: 325 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
composite of death and readmission | 30 days

SECONDARY OUTCOMES:
Correlation of MDW with SOFA and other sepsis markers (lactate, PVI, and procalcitonin) | 01 day

CONTACTS AND LOCATIONS:
Locations (1):
- Sahloul University Hospital, Sousse, Tunisia

IPD SHARING:
Plan to Share IPD: No